CLINICAL TRIAL: NCT00285974
Title: Dosage of Metal Ions in the Blood of Different Metal-on-metal Prostheses, in Correlation With Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003/398
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hip prosthesis (Experimental)
  Interventions: Device: metal-on-metal total hip prosthesis versus ceramic-on-ceramic total hip prosthesis

INTERVENTIONS:
Device: metal-on-metal total hip prosthesis versus ceramic-on-ceramic total hip prosthesis — metal-on-metal total hip prosthesis versus ceramic-on-ceramic total hip prosthesis

SUMMARY:
Prospective study including 6 groups of 20 patients with a total hip prosthesis. Five different types of metal-on-metal prostheses are studied, and 1 group with ceramic-on-ceramic prostheses acts as control group. Patients undergo a clinical evaluation and blood sampling preoperatively, and 3, 6, 12 and 24 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Hip osteoarthritis

Exclusion Criteria:

-

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2003-12 (Actual); Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Concentration of metal ions in the blood | preoperatively, and 3, 6, 12 and 24 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be